CLINICAL TRIAL: NCT01994213
Title: A Randomized, Single-arm, Open-label, Multicenter, Phase II Study of Famitinib as First/Second Line Treatment in Patients With Advanced or Metastatic Gastroenteropancreatic Neuroendocrine Tumor
Brief Title: A Study of Famitinib in Patients With Advanced or Metastatic Gastroenteropancreatic Neuroendocrine Tumor
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The applicant decided to close the study
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMTN- Ⅱ- GEPNET
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2013-11

CONDITIONS: Gastroenteropancreatic Neuroendocrine Tumor
Keywords: Famitinib; Gastroenteropancreatic Neuroendocrine Tumor; GEPNET
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor | interventions — famitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Famitinib (Experimental): Famitinib 25 mg qd p.o., 4 weeks per cycle.The treatment continued until disease progression or intolerable toxicity happened or patients withdrawal of consent.
  Interventions: Drug: Famitinib

INTERVENTIONS:
Drug: Famitinib — Famitinib 25 mg p.o. qd

SUMMARY:
Famitinib is a tyrosin-inhibitor agent targeting at c-Kit, VEGFR2, PDGFR, VEGFR3, Flt1 and Flt3. Phase I study has shown that the toxicity is manageable.

The purpose of this study is to evaluate the efficacy and safety profile of Famitinib in patients with advanced or metastatic Gastroenteropancreatic Neuroendocrine Tumor.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable advanced or metastatic, histologically-confirmed, gastroenteropancreatic neuroendocrine tumor. Tumors must be considered well-differentiated grade G1 or grade G2 in accordance with WHO 2010 classification.
* Must have at least one measurable disease by RECIST1.1 criteria(tumour lesions ≥10mm in longest diameter, malignant lymph nodes ≥15mm in short axis, scanning layer ≤ 5 mm).
* First-line therapy or second-line treatment (second-line treatment i.e. chemotherapy or cytokine therapy as first-line treatment failure or resistant patients).
* No previously received targeted therapy of gastroenteropancreatic neuroendocrine tumor (such as everolimus, sunitinib, or other tyrosine kinase or VEGF inhibitor treatment).
* Age between 18 and 75 years.
* ECOG Performance status ≤ 1.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with small-cell carcinoma, pheochromocytoma, paraganglioma or Merkel cell carcinoma
* Past or suffering from other cancer, but other than cure basal cell carcinoma and cervical carcinoma in situ
* Participated in other clinical trials within four weeks
* Concurrent therapy with somatostatin analogs(such as octreotide, lanreotide,etc.)
* A variety of factors that affect the oral medication (such as inability to swallow, gastrointestinal resection, chronic diarrhea and intestinal obstruction)
* Known brain metastases, spinal cord compression, cancer, meningitis, or screening CT or MRI examination revealed brain or leptomeningeal disease
* Subjects received surgery, chemotherapy, radiation therapy, cytokines treatment caused the damage has not been restored, the time interval ≤ 4 weeks, and the wound has not completely healed
* Participants have inadequate organ and marrow function as defined below:

  * hemoglobin < 90g/L
  * platelets < 100×10^9/L
  * neutrophils < 1.5×10^9/L
  * total bilirubin ≥ 1.25×ULN
  * serum transaminase(ALT and AST ) ≥ 1.5×ULN (If liver metastases are present, serum transaminase≥ 2.5×ULN)
  * creatinine clearance rate ≤ 60ml/min
  * cholesterol ≥ 1.5×ULN and triglyceride≥ 2.5 x ULN,
  * LVEF: < 50% by Color Doppler Ultrasonography
* Patients with uncontrollable hypertension after using single agent therapy (systolic blood pressure> 140 mmHg, diastolic blood pressure> 90 mmHg). Patients with more than Class I, myocardial ischemia or myocardial infarction, arrhythmia (including QT interval ≥ 450ms for male and 470ms for female) and class I heart failure.
* Urine protein ≥ + + and confirmed the 24-hour urinary protein>1.0 g
* Long-term untreated wounds or fractures
* Coagulopathy with bleeding tendency (such as active peptic ulcer)
* Previous artery / venous thromboembolic events, such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis and pulmonary embolism
* Application of anticoagulants or vitamin K antagonists such as warfarin, heparin or its analogues; If the prothrombin time international normalized ratio (INR) ≤ 1.5, with the purpose of prevention, the use of small doses of warfarin (1mg orally, once daily) or low-dose aspirin (less than 100mg daily) is allowed
* Female: All subjects who are not surgically sterile or postmenopausal must agree and commit to the use of a reliable method of birth control for the duration of the study and for 6 months after the last dose of test article. Child bearing potential, a negative urine or serum pregnancy test result before initiating Famitinib. Male: All subjects who are not surgically sterile or postmenopausal must agree and commit to the use of a reliable method of birth control for the duration of the study and for 6 months after the last dose of test article.
* Preexisting thyroid dysfunction, even using medical therapy, thyroid function cannot maintain in the normal range
* Abuse of psychiatric drugs or dysphrenia
* Immunodeficiency: HIV positive, or other acquired immunodeficiency, congenital immunodeficiency, or organ transplantation
* Evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | 12 weeks

SECONDARY OUTCOMES:
Progress free survival (PFS) | 3 years
Disease Control Rate (DCR) | 3 years
Overall Survival (OS) | 3 years
Quality of Life | 28-day cycle visit until disease progress
Percent of Participants with OS of one year | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jinwan Wang, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China